CLINICAL TRIAL: NCT03047798
Title: Comparative Effects of Aqueous Single-phase and Oil-water Two-phase Mouthrinses Containing Bamboo Salt, Magnolia Bark and Centella Asiatica Extracts on Reducing Gingivitis: a Randomized Clinical Trial
Brief Title: The Effect of Mouthrinses Containing Bamboo Salt, Magnolia Bark and Centella Asiatica on Reducing Plaque and Gingivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University (Other)
Collaborators: LG Household & Healthcare Ltd. (Unknown)
Responsible Party: Principal Investigator, Seungjae Choi, Dr. Resident, Seoul National University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S-D20140046
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Gingivitis; Dental Plaque
Keywords: centella asiatica; bamboo salt; magnolia bark; gingivitis; dental plaque; mouthrinse
MeSH Terms: conditions — Gingivitis; Dental Plaque

STUDY DESIGN:
Intervention Model Description: Subjects were instructed to use the prescribed mouthrinse to gargle their mouth for one minute, twice daily for two weeks. The completion of each experiment regimen was followed by a 2-week washout period, after which the subjects of each group were permutated to the next mouthrinse trial until all three groups underwent the three mouthrinse trial regimen.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The experiment was carried out in double-blind manner for the subjects and the examiner by providing the mouthrinses in opaque white bottles, labeled "A", "B" and "C".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aqueous single-phase mouthrinse (Experimental): This contained sodium fluoride and the additional ingredients of bamboo salt, magnolia bark and centella asiatica extracts in aqueous single-phase form.
  Interventions: Drug: Mouthrinse
- oil-water two-phase mouthrinse (Experimental): This contained sodium fluoride and the additional ingredients of bamboo salt, magnolia bark and centella asiatica extracts in oil-water two-phase form.
  Interventions: Drug: Mouthrinse
- Control (Placebo Comparator): The control mouthrinse only contained sodium fluoride
  Interventions: Drug: Mouthrinse

INTERVENTIONS:
Drug: Mouthrinse — A randomized clinical intervention study was planned with a cross-over design. The 34 subjects were randomly allocated to one of the three experimental groups: 1) the control; 2) ASM group for aqueous single-phase mouthrinse; 3) OTM group for oil-water two-phase mouthrinse.
  Subjects were instructed to use the prescribed mouthrinse to gargle their mouth for one minute, twice daily for two weeks. The completion of each experiment regimen was followed by a 2-week washout period, after which the subjects of each group were permutated to the next mouthrinse trial until all three groups underwent the three mouthrinse trial regimen.

SUMMARY:
This study aims to evaluate the effect of novel mouthrinse formulations containing bamboo salt, magnolia bark and centella asiatica extracts on gingivitis and dental plaque. Participants uses mouthrinses which contain bamboo salt, magnolia bark and centella asiatica extracts and the same participants will also use placebo for tooth brushing by cross-over design.

DETAILED DESCRIPTION:
This is a randomized clinical intervention study with a cross-over design. The subjects are randomly allocated to one of the three experimental groups: 1) the control; 2) ASM group for aqueous single-phase mouthrinse; 3) OTM group for oil-water two-phase mouthrinse. The experimental mouthrinses all contain sodium fluoride and the ASM and OTM contain additional ingredients of bamboo salt, magnolia bark and centella asiatica extracts. For the OTM, 50% essential oil is added to create an oil-water two-phase mouthrinse. Subjects are instructed to use the prescribed mouthrinse to gargle their mouth for one minute, twice daily for two weeks. The completion of each experiment regimen is followed by a 2-week washout period, after which the subjects of each group were permutated to the next mouthrinse trial until all three groups underwent the three mouthrinse trial regimen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults with at least 20 natural permanent teeth
* mild to moderate plaque (≥20% O'Leary index)
* mild gingivitis (20-30% BOP rate).

Exclusion Criteria:

* individuals undergoing orthodontic treatment
* individuals having deep periodontal pockets (≥ 6mm at two or more teeth) on more than two teeth
* diabetics
* pregnant or lactating women
* individuals taking antibiotics within the past one month
* individuals who have used any mouthwashes for the past 6 months.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2014-10-31 (Actual)

PRIMARY OUTCOMES:
Gingivitis | two weeks
  Gingival index
Dental plaque | two weeks
  Plaque index

IPD SHARING:
Plan to Share IPD: No